CLINICAL TRIAL: NCT05364190
Title: Efficacy and Safety of Early Initiation of Canagliflozin in Patients With Acute Decompansted Heart Failure
Brief Title: Canagliflozin in Patients With Acute Decompansted Heart Failure
Acronym: The CANA -AHF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: October 6 University (Other)
Collaborators: Cairo University (Other); National Heart Institute, Egypt (Other Government)
Responsible Party: Principal Investigator, rabab ahmed mohamed, Assistant lecturer ,MSc, October 6 University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL (2973)
Record Dates: First submitted 2022-04-25; First posted 2022-05-06 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Chronic Heart Failure; Acute Heart Failure; Diabetes Mellitus
Keywords: Canagliflozin; Hospitalized heart failure patients; I.V loop diuretic; NT-proBNP
MeSH Terms: conditions — Diabetes Mellitus | interventions — Canagliflozin; empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A(Intervention group) (Experimental): patients will receive 100 mg canagliflozin initiated within 24 hours from patients hospital admission due to signs of hypervolemic state. All patients also will be prescribed the conventional diuretic therapy and other medications such as angiotensin-converting enzyme inhibitors (ACEIs), angiotensin receptor blockers (ARBs), beta-blockers, angiotensin receptor-neprilysin inhibitor (ARNI) and mineralocorticoid receptor antagonists (MRAs). Canagliflozin will be continued for 90 days after hospital discharge
  Interventions: Drug: Canagliflozin
- Group B (Active Comparator): patients will receive 10 mg Empagliflozin initiated within 24 hours from patients hospital admission due to signs of a hypervolemic state.All patients also will be prescribed conventional diuretic therapy and other medications including ACEIs, ARBs, beta-blockers, ARNI, and MRAs.Empagliflozin will be continued for 90 days after hospital discharge
  Interventions: Drug: Empagliflozin

INTERVENTIONS:
Drug: Canagliflozin — Canagliflozin will be used in hospitalized heart failure patients regardless of their diabetic state.
  Arms: Group A(Intervention group)
Drug: Empagliflozin — Empagliflozin will be used in hospitalized heart failure patients regardless of their diabetic state.
  Arms: Group B

SUMMARY:
The study aims to investigate the efficacy and safety of the early initiation of canagliflozin treatment in hospitalized heart failure patients with volume overload (warm-wet) who require the use of I.V loop diuretic during the hospitalization period.

DETAILED DESCRIPTION:
The study will focus on the role of adding canagliflozin to I.V loop diuretic therapy early in unstable hospitalized acute heart failure patients regardless of diabetic state, patients who will be included in the study will continue on canagliflozin for 3 months after hospital discharge to evaluate the incidence of re-hospitalization, mortality rate and other benefits related to HF symptoms will be investigated.

ELIGIBILITY:
Inclusion Criteria:

Randomized within 24 of presentation during hospital admission for hypervolemic ADHF with evidence of congestion defined by the presence of any of the following signs or symptoms:

Peripheral edema Ascites Jugular venous pressure > 10 mmHg Orthopnea Paroxysmal nocturnal dyspnea 2.5 kg weight gain Signs of congestion on chest X-ray or lung ultrasound If pulmonary artery catheterization is available pulmonary capillary wedge pressure > 19 mmHg plus a systemic physical examination finding of hypervolemia.

Planned use of intravenous (IV) loop diuretic therapy during the current hospitalization Estimated glomerular filtration rate (e-GFR) > 30 mL/min/1.73 m2 based on the Modification of Diet in Renal Disease (MDRD) equation.

Exclusion Criteria:

Type 1 diabetes Serum glucose < 80 mg/dL Systolic blood pressure < 90 mmHg Requirement of IV inotropic therapy History of hypersensitivity to any SGLT-2 inhibitors Already receiving therapy with an SGLT2 inhibitor Women who are pregnant or breastfeeding Severe anemia (Hemoglobin < 7.5 g/dL)(24) Severe uncorrected aortic or mitral stenosis Inability to perform standing weights or measure urine output accurately Signs of ketoacidosis and/or hyperosmolar hyperglycaemic syndrome (pH >7.3 and glucose > 250 mg/dL and HCO3 > 18 mmol/L) in diabetic patients at the time of inclusion to the study.

The use of other diuretic therapies including; ≥100 mg/day spironolactone doses, ≥ 100 mg/day eplerenone, metolazone, hydrochlorothiazide, or other thiazides, systemic acetazolamide for the indication of diuretics, triamterene, or amiloride therapy.

The use of other medications possessing natriuretic effect as nesiritide, or arginine vasopressin antagonists.

Diffuse anasarca with 4+ edema and projected hypervolemia exceeding 18 kg. Severe hepatic impairment (Child-Pugh class C). Patients on hemodialysis Acute myocardial infarction with symptoms of acute ischemia or changes on electrocardiogram

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2022-06-04 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
The cumulative mean of daily diuresis | After (day1)24 hours from hospital admission and until Day 5 or discharge if earlier
  which is define as total urine output in 24 hours during the hospitalization period.

SECONDARY OUTCOMES:
Measuring diuretic response | Baseline to hospital discharge, an average of 5-6 days
  which is the cumulative change in weight (kg) from enrollment until discharge adjusted for cumulative diuretic dose in IV furosemide or equivalents
The change in the level of NT-pro BNP | Baseline to hospital discharge, an average of 5-6 days
  The change in the level of NT-pro BNP between the hospital admission day and the day of discharge.
Presence of symptoms of congestion and dyspnea at discharge | Baseline to hospital discharge, an average of 5-6 days.
  measured via the change in visual analogue scale (VAS) dyspnea score between enrollment day and the discharge day. the score goes between 0-10 where 0 = no breathlessness to 10 = worst breathlessness possible.
Intensive care unit (ICU) length of stay | Baseline to hospital discharge, an average of 5-6 days
  measured as days from admission to ICU to discharge.
The incidence of worsening of heart failure case | Baseline to hospital discharge, an average of 5-6 days.
  which is defined as failure of IV diuretic regimen to stabilize the patient state during hospitalization which requires the use of IV inotropic therapy
Fractional Excretion of Sodium (FENa)-based diuretic efficiency | Baseline to hospital discharge, an average of 5-6 days.
  FENa per 40 mg of IV furosemide equivalents of loop dose using spot urine collected 24 hours after continues infusion of loop dose beginning and every day until patients discharge from hospital.
Serum potassium | Baseline to hospital discharge, an average of 5-6 days.
  Serum potassium covariate with attention to both elevation and depression on a daily basis during hospitalization period.
Incidence of ketoacidosis | Baseline to 90 days post discharge
  reporting ketoacidosis
Serum glucose covariate adjusted for baseline with attention to both elevation | Baseline to hospital discharge, an average of 5-6 days.
  (> 400 mg/dL) and depression (< 70 mg/dL).
Incidence of symptomatic, sustained hypovolemic hypotension | Baseline to hospital discharge, an average of 5-6 days.
  systolic blood pressure < 90 mmHg over 30 minutes requiring fluid administration
In-hospital mortality | Baseline to hospital discharge, an average of 5-6 days.
  incidence of mortality
Hospital readmission within 90 days of discharge for heart failure | within 90 post discharge
  Re-hospitalization within 90 days from hospital discharge
Incidence of mortality within 90 days from discharge due cardiovascular cause | within 90 post discharge
  Incidence of mortality
The incidence of worsening of renal function | Baseline to 90 post discharge
  which is defined as a decline in the e-GFR of 50% or greater from the baseline during any follow-up points
Any reported adverse events during follow up period. | within 90 post discharge
  ketoacidosis, genital mycotic infection, urinary tract infection, Fournier's gangrene, fractures, or amputation
The progression of heart failure severity | within 90 post discharge
  via measuring Kansas City Cardiomyopathy Questionnaire - Total Symptom Score (KCCQ-TSS)
  .all KCCQ scores are scaled from 0 to 100 and frequently summarized in 25-point ranges, where scores represent health status as follows: 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; and 75 to 100: good to excellent

CONTACTS AND LOCATIONS:
Locations (1):
- National heart institute, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The study results will be duplicated after the end of the study
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 2024